CLINICAL TRIAL: NCT07351968
Title: A Multicenter, Randomized, Double-blind, Agent-positive and Placebo-controlled, Parallel-group Phase Ib Study to Evaluate the Efficacy and Safety of HRS-2129 in Patients With Knee Osteoarthritis
Brief Title: A Phase Ib Study to Evaluate the Efficacy and Safety of HRS-2129 in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2129-106
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Moderate Pain in Knee Osteoarthritis; Severe Pain in Knee Osteoarthritis
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: Comparison between HRS-2129 high dose group, HRS-2129 low dose group, Celecoxib positive control group, and Placebo control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HRS-2129 High Dose Group (Experimental): HRS-2129 high dose group.
  Interventions: Drug: HRS-2129 Tablet; Drug: Celecoxib Capsule Placebo; Drug: HRS-2129 Tablet Placebo
- HRS-2129 Low Dose Group (Experimental): HRS-2129 low dose group.
  Interventions: Drug: HRS-2129 Tablet; Drug: Celecoxib Capsule Placebo; Drug: HRS-2129 Tablet Placebo
- Celecoxib Group (Active Comparator): Celecoxib group.
  Interventions: Drug: Celecoxib capsule; Drug: HRS-2129 Tablet Placebo
- Placebo Group (Placebo Comparator): Placebo group.
  Interventions: Drug: Celecoxib Capsule Placebo; Drug: HRS-2129 Tablet Placebo

INTERVENTIONS:
Drug: HRS-2129 Tablet — HRS-2129 tablet.
  Arms: HRS-2129 High Dose Group; HRS-2129 Low Dose Group
Drug: Celecoxib capsule — Celecoxib capsule.
  Arms: Celecoxib Group
Drug: Celecoxib Capsule Placebo — Celecoxib capsule placebo.
  Arms: HRS-2129 High Dose Group; HRS-2129 Low Dose Group; Placebo Group
Drug: HRS-2129 Tablet Placebo — HRS-2129 tablet placebo.

SUMMARY:
Primary Objective: To explore the effectiveness of different doses of HRS-2129 in the treatment of patients with moderate to severe pain in knee osteoarthritis. Secondary Objectives: To evaluate the safety of different doses of HRS-2129 for the treatment of patients with moderate to severe pain in knee osteoarthritis; To evaluate the population pharmacokinetic profile of HRS-2129 in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before starting the activities related to the trial;
2. The Numerical Evaluation Scale (NRS) pain score of the index knee joint at screening is ≥ 4;
3. Subjects must be willing to discontinue all medical and non-medical treatments for osteoarthritis pain except rescue medication (acetaminophen) and not use prohibited analgesics throughout the study ;
4. Male and female subjects of childbearing potential must agree to use highly effective contraceptive measures with their partners from the signing of the informed consent form until 1 month after the last dose of investigational product.

Exclusion Criteria:

1. History of other diseases that may involve the target joint;
2. History of major trauma or surgery of knee joint and hip joint in the past year;
3. Plan to undergo surgical procedure during the study;
4. Most or complete loss of mobility;
5. There are other diseases that may confuse the assessment of osteoarthritis pain;
6. There is a neuropsychiatric disease, and the investigator's assessment may affect the evaluation of osteoarthritis (OA) or self-score;
7. There are serious or poorly controlled concomitant diseases;
8. Those who have a clear history of peptic ulcer, bleeding, perforation or obstruction within 1 year before screening, and have been clinically diagnosed;
9. Those who require drug treatment or surgical intervention;
10. History of malignant tumors within 5 years before screening;
11. Have a history of drug abuse, drug abuse and/or alcoholism within 2 years before screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale scores. | At week 4.

SECONDARY OUTCOMES:
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale scores. | From baseline to Week 1, 2 and 3.
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) joint function subscale scores. | From baseline to Week 1, 2, 3 and 4.
Change from baseline in the weekly mean (Week 1, 2, 3 and 4) of the index Knee Numerical Rating Scale (NRS) pain score (resting). | From baseline to Week 1, 2, 3 and 4.
Change from baseline in the weekly mean (Week 1, 2, 3 and 4) of the index Knee Numerical Rating Scale (NRS) pain score (flat walking). | From baseline to Week 1, 2, 3 and 4.
Change from baseline in the overall patient global assessment (PGA) of osteoarthritis condition using the 5-point Likert scale. | From baseline to Week 1, 2, 3 and 4.
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness subscale scores. | From baseline to Week 1, 2, 3 and 4.
Change from baseline in total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. | From baseline to Week 1, 2, 3 and 4.
Treatment response: WOMAC pain subscale scores decreased by ≥ 30%, ≥ 50%, ≥ 70% from baseline. | At Week 1, 2, 3 and 4.
Adverse events (AEs) occurred during the study. | During the study, approximately 8 months.
  To evaluate the safety and tolerability of HRS-2129 tablets.
Serious adverse events (SAEs) occurred during the study. | During the study, approximately 8 months.
  To evaluate the safety and tolerability of HRS-2129 tablets.

CONTACTS AND LOCATIONS:
Locations (1):
- Drum Tower Hospital affiliated to Nanjing University School of Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided